CLINICAL TRIAL: NCT00737256
Title: A Double-Blind, Controlled Study of Aripiprazole in Co-Morbid Schizophrenia and Cocaine Dependence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul Saenger (Other)
Responsible Party: Sponsor-Investigator, Paul Saenger, Executive Director, Denver Research Institute
Organization: Denver Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-0124; NCT00819689 (obsolete NCT alias)
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia; Cocaine Dependence
MeSH Terms: conditions — Schizophrenia; Cocaine-Related Disorders | interventions — Aripiprazole; Perphenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Aripiprazole
- 2 (Active Comparator)
  Interventions: Drug: Perphenazine

INTERVENTIONS:
Drug: Aripiprazole — 15-30 mg
  Arms: 1
Drug: Perphenazine — 8-16 mg
  Arms: 2

SUMMARY:
The purpose of this study is to gather systematic clinical data on whether aripiprazole, a partial dopamine agonist, beneficially affects schizophrenia plus cocaine dependence subjects. Since aripiprazole has established effects against schizophrenia, the study focuses on whether aripiprazole concurrently reduces co-morbid cocaine dependence in schizophrenia plus cocaine dependence sufferers compared to a standard typical antipsychotic treatment (perphenazine). The working hypothesis states that subjects in the aripiprazole treatment arm of the study will give fewer cocaine positive urine specimens as compared to the perphenazine control arm.

ELIGIBILITY:
Inclusion Criteria:

1. Have a primary DSM-IV diagnosis of Schizophrenia or Schizoaffective disorder
2. Have a DSM-IV diagnosis of current cocaine dependence.
3. Are capable of reading, comprehending, and signing informed consent.
4. Agree to take Aripiprazole or Perphenazine as treatment for SCHZ and CD.
5. Agree to stop taking any other antipsychotic medication
6. If female and of child bearing potential (WOCBP) agree to use an acceptable form of birth control and have a negative pregnancy test within 2 days prior to starting study medication

Exclusion Criteria:

1. Under 18 years old or over 65 years old.
2. Refusal or inability to give informed consent,
3. Have a history of myocardial infarction or ischemic heart disease, heart failure or conduction abnormalities, cerebrovascular disease, or conditions that would predispose to hypotension (dehydration, hypovolemia),
4. A history of seizures or conditions that lower the seizure threshold
5. Have current suicidal ideation (history of suicide attempt in past 60 days)
6. Are actively psychotic which in the opinion of the investigator would preclude proper informed consenting or protocol adherence
7. Are receiving or plan to receive an agent metabolized by the Cytochrome P450-3A4 or -2D6 systems, including carbamazepine, ketoconazole, quinidine, fluoxetine, and paroxetine
8. WOCBP not on, or do not agree to use an acceptable form of contraception
9. Known sensitivity to aripiprazole or perphenazine
10. A diagnosis of current or past tardive dyskinesia
11. Pending legal charges or a court mandate for drug treatment
12. Currently taking concomitant medications that have been shown to reduce cocaine use, such as disulfiram
13. Clinically significant liver function abnormalities
14. Currently receiving depot neuroleptics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of negative urine drug screen results will be significantly greater in the subjects treated with aripiprazole than in those treated with perphenazine. | Week 3 and Week 8 of study participation

SECONDARY OUTCOMES:
The mean total self-report cocaine use days will be significantly fewer in subjects treated with aripiprazole than in those treated with perphenazine. | End of study participation
The mean cocaine craving scores will be lower in subjects treated with aripiprazole than in those treated with perphenazine. | End of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Beresford, MD, Principal Investigator — Denver Veteran's Affairs Medical Center
Locations (1):
- Veteran's Affairs Medical Center, Denver, Colorado, United States